CLINICAL TRIAL: NCT07026175
Title: Unravelling Energy Issues Underpinning Low Energy Availability in High Performance Athletes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Australian Catholic University (Other)
Collaborators: Wu Tsai Human Performance Alliance (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-4078HC
Record Dates: First submitted 2025-05-28; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Relative Energy Deficiency in Sport
Keywords: Relative Energy Deficiency in Sport (REDs); Endurance; Athlete; Sleeping Metabolic Rate; Problematic Low Energy Availability
MeSH Terms: conditions — Relative Energy Deficiency in Sport

STUDY DESIGN:
Intervention Model Description: This project employs a nonblinded three-sequence crossover design. All participants will undertake a control trial followed by a counterbalanced allocation to one of the low energy availability (LEA) trials, then they will complete the other low energy availability trial. All trials will have a minimum 3-week washout period between them. Allocation to the LEA trials will be randomised and stratified for sex.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Trial (No Intervention): A 6-day control trial. All participants will commence with this trial involving an energy availability of 40 kcal/kg fat-free mass (FFM). Energy intake will be 55 kcal/kg FFM/d and exercise energy expenditure will be 15 kcal/kg FFM/d. This will be followed by a minimum 3-week washout period where the participant will be advised to return to their routine diet and exercise.
- Low Energy Availability - Diet (Experimental): A 6-day severe low energy availability (LEA, 15kcal/kg FFM/d) trial, achieved by superimposing restricted energy intake on the HEA trial. Energy intake will be 30 kcal/kg FFM/d and exercise energy expenditure will be 15 kcal/kg FFM/d. This will be followed by a minimum 3-week washout period where the participant will be advised to return to their routine diet and exercise.
  Interventions: Other: Diet-induced low energy availability
- Low Energy Availability - Exercise (Experimental): A 6-day severe low energy availability (LEA, 15kcal/kg FFM/d) trial, achieved by superimposing increased exercise energy expenditure on the HEA trial. Energy intake will be 45 kcal/kg FFM/d and exercise energy expenditure will be 30 kcal/kg FFM/d. This will be followed by a minimum 3-week washout period where the participant will be advised to return to their routine diet and exercise.
  Interventions: Other: Exercise-induced low energy availability

INTERVENTIONS:
Other: Diet-induced low energy availability — 6-days of severe low energy availability (LEA, 15kcal/kg FFM/d), achieved by superimposing restricted energy intake on the control trial.
  Arms: Low Energy Availability - Diet
Other: Exercise-induced low energy availability — 6-days of severe low energy availability (LEA, 15kcal/kg FFM/d), achieved by superimposing increased exercise energy expenditure on the control trial.
  Arms: Low Energy Availability - Exercise

SUMMARY:
The goal of this clinical trial is to understand how the body responds to short-term, severe low energy availability (LEA) in healthy, weight-bearing endurance athletes aged 18-45 years old. LEA describes a mismatch between an individual's dietary energy intake and the energy cost of their commitments for training and competition. The main questions this trial aims to answer are:

1. What effect does short-term, severe LEA have on sleeping metabolic rate?
2. What effect does short-term, severe LEA have on other body systems identified within the Relative Energy Deficiency in Sport (REDs) Health and Performance Conceptual models?

Researchers will compare a control trial with both a LEA trial achieved through diet restriction and a LEA trial achieved through increased exercise to see if there are differences in the body's response.

Participants will complete three 6-day trials, a minimum of 3-weeks apart, involving:

* Prescribed diet (all food provided)
* Prescribed running and/or cycling exercise
* Two visits to ACU Fitzroy campus for blood tests and exercise testing
* 50 hour stay (two nights and two days) in the ACU metabolic chamber

DETAILED DESCRIPTION:
The study will involve a three-sequence crossover design, with participants undertaking a control trial first, involving energy availability of 40 kcal/kg fat free mass (FFM) and a 15 kcal/kg FFM exercise energy expenditure (EEE) as baseline training volume, before a counterbalanced allocation to low energy availability via dietary restriction (LEADIET) or low energy availability via increased exercise energy expenditure (LEAEX). This design will allow further screening of Relative Energy Deficiency in Sport (REDs) risk, identify participants who are likely to be unable to fulfil the exercise commitments of LEAEX and avoid the unknown carryover effects of two consecutive low energy availability (LEA) trials on the subsequent control trial, as would occur in some participants with a fully counterbalanced treatment allocation.

Baseline testing (body composition/bone mineral density via DXA, aerobic capacity, LEA hormone blood panel, vitamin D, resting metabolic rate, REDs screening via REDs-CAT2) will be undertaken to confirm inclusion and develop individualised diet and training plans. Thereafter, participants will undertake a 6-day supervised exposure to energy availability of ~40 kcal/kg FFM/d, involving supplied meals and prescribed daily running/race walking. For female participants, trials will commence within days 1-5 of the menstrual cycle, to ensure that all testing occurs in the same (follicular) phase. A minimum 3-week washout period will occur between trials, with participants being guided to return to habitual training and dietary habits. Trials 2 and 3 will consist of exposure to severe LEA (15 kcal/kg FFM/d), which is achieved either by superimposing restricted energy intake (EI) or increased (doubled) EEE on the previous training plan.

Diet plans and food provision will be managed by experienced sports dietitians to incorporate individual preferences and intolerances. While participants are free-living at the start of each trial week, food drops will be undertaken to check well-being and compliance to the diet/ training intervention. The final 2 days of residence at ACU facilities (medical unit and metabolic chamber) will allow more comprehensive data collection. Individual protocols (described briefly below) have been previously developed by our group and collaborators. Together, they will investigate within and between trial changes in metrics representing the range of body systems that have been identified at risk of perturbations due to LEA within the REDs Conceptual Health and Performance Models.

Summary of the protocols completed in this study:

1. VO2 max: Running protocol: Measured once at screening visit (and potentially remeasured if participant trials are spaced >3 months apart and aerobic fitness requires rechecking)
2. Resting Metabolic Rate: Outpatient protocol via Parvo metabolic cart: Measured once in baseline testing to enable calculation of EA components for intervention
3. DXA: total body composition: Measured once at screening visit to enable calculation of EA components for intervention, and twice in each trial (Day 1 and Day 5)
4. DXA: bone mineral density (Hip and Spine): Measured once at screening visit
5. Cognitive tests: 5-minute psychomotor vigilance test (PVT) & 3-minute Simon Squared, delivered via Inquisit software (screening visit, then Day 1 and Day 6)
6. RESTQ-76: questionnaire of overall wellbeing (Day 6)
7. Diet feedback questionnaire (Day 6)
8. Oura Ring: sleep characteristics, resting heart rate (HR), total energy expenditure (EE), basal body temperature, HR variability (HRV) (throughout each trial)
9. Somfit: sleep architecture (Night of Days 3, 4, and 5)
10. Training capacity: Garmin-derived HR and EE, rate of perceived exertion (RPE, throughout trial), metabolic, physiological and perceptual responses during standardised running test (Day 5)
11. Dietary iron absorption and incorporation: Intake of stable isotope (3.8mg, Fe57 as ferrous sulphate) (evening of Day 4), with 8 blood samples collected from 0-480 min post dose to assess iron absorption. A further blood sample taken after 28 days will measure incorporation into red blood cells to assess functional iron availability
12. Venepuncture/Venous cannulation: Total blood volume per trial = 140 ml for:

    * LEA panel: testosterone, estrogen, progesterone, IGF-1, T3, leptin, iron status, lipids, glucose/insulin (screening visit, Day 1 and Day 5)
    * Hormone pulsatility: 8 h @15 min collection of Luteinising Hormone, Growth Hormone, Cortisol (overnight Day 4)
    * Appetite peptides: Leptin, Active Ghrelin, PP, GLP-1, PYY (Day 5)
    * Immune response: IL-6, mitochondrial respiration, reactive oxygen species emission, and protein expression in peripheral blood mononuclear cells (PBMCs), circulating leukocyte type distribution and mobilisation, circulating cell-free DNA (Day 5)
    * Bone turnover: CTX-1 and P1NP (Day 5)
    * Iron absorption and response: plasma iron-isotope appearance (overnight Day 4), Hepcidin (Day 5)
13. Exercise metabolism: blood lactate, glucose (finger prick collection, Day 5 exercise)
14. Gut comfort: Standardised GI questionnaire pre- and post-exercise (Day 5 exercise)
15. Protein turnover: Consumption of stable isotopes of 15N-glycine and D3-3-methyl-histidine (Day 4), with a baseline urine sample, and serial timed samples (Days 5 and 6) will allow determination of whole-body protein turnover (measured as 15N-Alanine), and muscle proteolysis
16. Bone breakdown: Measurement of Ca isotope abundance in urine (on waking urine sample on Day 1 and 24-hour urine sample on Day 5/6 in metabolic chamber) will allow assessment of bone breakdown (periods of greater bone breakdown: formation will see greater abundance of lighter isotopes).
17. Metabolic chamber: 24 h energy expenditure, sleeping metabolic rate, basal metabolic rate, EEE (Day 5/6 in metabolic chamber)
18. Blood glucose monitoring: blood glucose monitoring, using continuous glucose monitors (Freestyle Libre Pro iQ) (from Day 1 through to end of Day 6)

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Well trained weight-bearing athlete (tier 2-4 1)
* Perform ~45km per week of weight-bearing endurance training, and able to undertake the prescribed exercise in each trial condition
* Pass the ESSA pre-exercise screening tool and/or obtain GP clearance to exercise

Exclusion Criteria:

* Assessment of red status on the REDs Clinical Assessment Tool
* Unable to attend ACU in Fitzroy, Victoria, for the 6 study visits for completion of the study protocol
* Pregnancy
* Use of hormonal contraceptive with the previous 3 months
* Onset of peri/menopause

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Sleeping metabolic rate between trials, measured using a human metabolic chamber on night 5 of each trial condition. | Night 5 of each trial condition from enrolment to the end of the third trial period.
  The primary outcome is the within-participant and sex-based difference in Sleeping Metabolic Rate (SMR) across the three trial conditions. Analyses will also compare differences in SMR responses between sexes.

OTHER OUTCOMES:
Fasting values of metabolic and reproductive hormones between trials. | Day 1 of each trial condition from enrollment to Day 5 of the third trial period.
  Within-participant and sex-based changes in fasting values of metabolic and reproductive hormones (testosterone, estrogen, progesterone, IGF-1, T3, leptin, iron status, lipids, glucose/insulin). Measured via venous blood sample on day 1 and day 5 of each trial.
Overnight pulsatility of luteinising hormone between trials. | Night 4 of each trial condition from enrolment to Day 5 of the third trial period.
  The secondary outcome is within-participant and sex-based difference in overnight pulsatility of luteinising hormone. This will be measured via venous blood samples taken every 15 minutes for 8 hours on night 4 of each trial.
Overnight pulsatility of growth hormone between trials. | Night 4 of each trial condition from enrolment to Day 5 of the third trial period.
  The secondary outcome is within-participant and sex-based difference in overnight pulsatility of growth hormone. This will be measured via venous blood samples taken every 15 minutes for 8 hours on night 4 of each trial.
Overnight pulsatility of cortisol between trials. | Night 4 of each trial condition from enrolment to Day 5 of the third trial period.
  The secondary outcome is within-participant and sex-based difference in overnight pulsatility of cortisol. This will be measured via venous blood samples taken every 15 minutes for 8 hours on night 4 of each trial.
Dietary iron absorption and regulation between trials. | Night 4 of each trial from enrolment, to 28 days post the third trial period.
  Within-participant and sex-based change in dietary iron absorption and regulation (plasma iron-isotope (Fe57) appearance), measured via blood sample collected 0-480minutes and at 28 days after intake of stable isotope Fe57.
Substrate utilisation during a standardised exercise protocol between trials. | Day 5 of each trial condition from enrolment to Day 5 of the third trial period.
  Within-participant and sex-based change in substrate utilisation, during a standardised exercise protocol between trials. This will be measured by venous and capillary blood samples on Day 5 of each trial.
Abundance of naturally occurring isotopes of calcium in urine between trials. | Days 1, 4, 5 and 6 of each trial condition from enrolment to Day 6 of the third trial period.
  Within-participant and sex-based change in abundance of naturally occurring isotopes of calcium (40Ca, 42Ca, 43Ca, 44Ca, 46Ca, and 48Ca) in urine, to predict boen metabolism. This will be measured via first void urine samples collected on days 1 and 4, and 24-hour urine collection on days 5-6 of each trial.
Immune markers between trials. | Day 5 of each trial, from enrolment to day 5 of the third trial period.
  Within-participant and sex-based difference in immune markers (IL-6, mitochondrial respiration, reactive oxygen species emission and protein expression in peripheral blood mononuclear cells (PBMCs), circulating leukocyte type distribution and mobilisation, circulating cell-free DNA). This will be measured via blood sample on day 5 of each trial.
Whole-body protein turnover and muscle proteolysis between trials. | Days 5-6 of each trial condition from enrolment to the end of the third trial period.
  Within-participant and sex-based difference in whole-body protein turnover (measured as 15N-Alanine) and muscle proteolysis. This will be measured via 24-hour urine collection on days 5-6.
Cognitive control between trials. | Days 1 and 6 of each trial condition from enrolment to day 6 of the third trial period.
  Within-participant and sex-based change in cognitive control assessed via the 3-minute Simon Squared, delivered via Inquisit software. This will be measured on days 1 and 6 of each trial.
Cognitive arousal between trials. | Days 1 and 6 of each trial condition from enrolment to day 6 of the third trial period.
  Within-participant and sex-based change in cognitive arousal, assessed via the 5 minute psychomotor vigilance test, delivered via Inquisit software. This will be measured on days 1 and 6 of each trial.
Semi-targeted lipidomics between trials. | Day 5 of each trial condition from enrolment to day 5 of the third trial period.
  Within participant and sex-based difference in lipidomics measured via venous blood sample on day 5 of each trial.
Interstitial fluid glucose levels between trials. | Days 1-6 of each trial condition from enrolment to the end of day 6 of the third trial period.
  Within-participant and sex-based difference of interstitial glucose levels between trials. This will be measured using continuous glucose monitors worn from day 1 to day 6 of each trial condition.
Duration of sleep stages between trials. | Nights 3-5 of each trial condition from enrolment to day 6 of the third trial period.
  Within-participant and sex-based difference in duration (minutes) of sleep stages per night on nights 3-5 of each trial period, measured using the Somfit wearable device.
Sleep quantity between trials. | Nights 1-5 of each trial condition from enrolment to day 6 of the third trial period.
  Within-participant and sex-based difference in sleep quantity (total sleep time) measured using the Oura Ring wearable device on nights 1-5 throughout the trial periods.
Sleep onset time between trials. | Nights 3-5 of each trial condition from enrolment to day 6 of the third trial period.
  Within-participant and sex-based difference in sleep onset time on nights 3-5 of each trial period, measured using the Somfit wearable device and Oura Ring.
Sleep offset time between trials. | Nights 3-5 of each trial condition from enrolment to day 6 of the third trial period.
  Within-participant and sex-based difference in sleep offset time on nights 3-5 of each trial period, measured using the Somfit wearable device and Oura Ring.
Sleep onset latency between trials. | Nights 3-5 of each trial condition from enrolment to day 6 of the third trial period.
  Within-participant and sex-based difference in sleep onset latency on nights 3-5 of each trial period, measured using the Somfit wearable device.
Rapid eye movement (REM) onset latency between trials. | Nights 3-5 of each trial condition from enrolment to day 6 of the third trial period.
  Within-participant and sex-based difference in REM onset latency on nights 3-5 of each trial period, measured using the Somfit wearable device.
Number of awakenings per night between trials. | Nights 3-5 of each trial condition from enrolment to day 6 of the third trial period.
  Within-participant and sex-based difference in number of awakenings per night on nights 3-5 of each trial period, measured using the Somfit wearable device.
Sleep quality between trials. | Nights 1-5 of each trial condition from enrolment to day 6 of the third trial period.
  Within-participant and sex-based difference in sleep quality (total sleep time as a percentage of time in bed) measured using the Oura Ring wearable device on nights 1-5 throughout the trial periods.

CONTACTS AND LOCATIONS:
Overall Officials: Louise M Burke, PhD, Principal Investigator — Australian Catholic University
Locations (1):
- Australian Catholic University, Fitzroy, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available from the corresponding author for a period of 36 months from publication, upon reasonable request for academic use. The data will not be made publicly available, as it contains information that could compromise research participant consent.
Time Frame: For a period of 36 months from publication of the primary outcome.

REFERENCES:
- [Background] Burke LM, Ackerman KE, Heikura IA, Hackney AC, Stellingwerff T. Mapping the complexities of Relative Energy Deficiency in Sport (REDs): development of a physiological model by a subgroup of the International Olympic Committee (IOC) Consensus on REDs. Br J Sports Med. 2023 Sep;57(17):1098-1108. doi: 10.1136/bjsports-2023-107335. PMID 37752007
- [Background] Mountjoy M, Ackerman KE, Bailey DM, Burke LM, Constantini N, Hackney AC, Heikura IA, Melin A, Pensgaard AM, Stellingwerff T, Sundgot-Borgen JK, Torstveit MK, Jacobsen AU, Verhagen E, Budgett R, Engebretsen L, Erdener U. 2023 International Olympic Committee's (IOC) consensus statement on Relative Energy Deficiency in Sport (REDs). Br J Sports Med. 2023 Sep;57(17):1073-1097. doi: 10.1136/bjsports-2023-106994. PMID 37752011
- [Background] Loucks AB, Kiens B, Wright HH. Energy availability in athletes. J Sports Sci. 2011;29 Suppl 1:S7-15. doi: 10.1080/02640414.2011.588958. Epub 2011 Jul 28. PMID 21793767